CLINICAL TRIAL: NCT01708902
Title: A Phase III Randomised, Double-blind, Double-dummy, Parallel Group Study to Compare the Efficacy and Safety of Twice Daily Administration of the Fix Dose Combination of Linagliptin 2.5 mg + Metformin 500 mg, or of Linagliptin 2.5 mg + Metformin 1000 mg, With the Individual Components of Metformin (500 mg or 1000 mg, Twice Daily), and Linagliptin (5.0 mg, Once Daily) Over 24 Weeks in Treatment naïve Type 2 Diabetic Patients With Insufficient Glycaemic Control
Brief Title: Study to Compare the Efficacy and Safety of Administration of the Fix Dose Combination of Linagliptin Plus Metformin in Drug naïve Type 2 Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1288.18
Record Dates: First submitted 2012-10-16; First posted 2012-10-17 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; Metformin

ARMS (5):
- linagliptin2.5mg / metformin500mg BID (Experimental): patient to receive a tablet containing linagliptin 2.5mg and metformin 500mg BID
  Interventions: Drug: linagliptin 5mg; Drug: Metformin 500mg
- linagliptin2.5mg / metformin1000mg BID (Experimental): patient to receive a tablet containing linagliptin 2.5mg and metformin 1000mg BID
  Interventions: Drug: linagliptin 5mg; Drug: Metformin 1000mg
- metformin 500mg BID (Active Comparator): patient to receive a tablet containing metformin 500mg BID
  Interventions: Drug: linagliptin2.5mg/metformin500mg
- metformin 1000mg BID (Active Comparator): patient to receive a tablet containing metformin 1000mg BID
  Interventions: Drug: linagliptin2.5mg/metformin1000mg
- linagliptin 5 mg QD (Active Comparator): patient to receive a tablet containing linagliptin 5mg once daily
  Interventions: Drug: linagliptin2.5mg/metformin1000mg; Drug: linagliptin2.5mg/metformin500mg

INTERVENTIONS:
Drug: linagliptin2.5mg/metformin1000mg — linagliptin2.5mg/metformin1000mg BID
  Arms: metformin 1000mg BID
Drug: linagliptin2.5mg/metformin1000mg — linagliptin2.5mg/metformin1000mg BID
  Arms: linagliptin 5 mg QD
Drug: linagliptin 5mg — linagliptin 5mg once daily
  Arms: linagliptin2.5mg / metformin500mg BID
Drug: Metformin 500mg — Metformin 500mg BID
  Arms: linagliptin2.5mg / metformin500mg BID
Drug: linagliptin2.5mg/metformin500mg — linagliptin2.5mg/metformin500mg BID
  Arms: metformin 500mg BID
Drug: linagliptin2.5mg/metformin500mg — linagliptin2.5mg/metformin500mg BID
  Arms: linagliptin 5 mg QD
Drug: linagliptin 5mg — linagliptin 5mg once daily
  Arms: linagliptin2.5mg / metformin1000mg BID
Drug: Metformin 1000mg — Metformin 1000mg BID
  Arms: linagliptin2.5mg / metformin1000mg BID

SUMMARY:
Reduced factorial design study with 24 week randomized treatment of initial combination therapy with linagliptin and metformin in T2DM patients

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of Type 2 diabetes mellitus(T2DM) prior to informed consent
2. Male and female patients on diet and exercise regimen who are drug-naïve
3. Glycosylated haemoglobin A1c (HbA1c) at V1a >/=7.5 %<11% for main group and HbA1c >/= 11.0 % for the additional parallel group
4. Age >/= 18 and </= 80 years at Visit 1a (Screening)
5. Body Mass Index(BMI)</ = 40 kg/m2 at Visit 1a (Screening)
6. Signed and dated written informed consent by date of Visit 1a in accordance with good clinical practice(GCP) and local legislation

Exclusion criteria:

1. Uncontrolled hyperglycaemia required for rescue medication during placebo run-in phase
2. In main group, the patients with investigational medicinal product(IMP) compliance < 80 % or >120 % during 2 weeks placebo run in period
3. Acute coronary syndrome stroke or Transient ischaemic attack (TIA) within 3 months prior to randomisation
4. Impaired hepatic function, defined by serum levels of either Alanine aminotransferase(ALT) ,Aspartate aminotransferase(AST), or alkaline phosphatase (AP) above 3 x upper limit of normal (ULN) ,or total bilirubin above 1.5 x ULN as determined at Visit 1a
5. Known hypersensitivity or allergy to linagliptin or its excipients or metformin or placebo
6. Treatment with anti-obesity drugs 3 months prior to informed consent or any other treatment at the time of screening
7. Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake in the opinion of the investigator.
8. Concurrent participation in another clinical trial or any investigational therapy within thirty days prior to signing the consent form or during the trial.
9. Pre-menopausal women (last menstruation </= 1 year prior to informed consent) who are nursing or pregnant or are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study
10. Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent.
11. Renal failure or renal impairment at Visit 1a (screening) with an Estimated Glomerular Filtration Rate(eGFR) < 60 ml/min
12. Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption
13. Dehydration by clinical judgement of the investigator
14. Clinical detected unstable or acute congestive heart failure
15. Acute or chronic metabolic acidosis (present in patient history)
16. Hereditary galactose intolerance
17. Known history of pancreatitis and chronic pancreatitis
18. Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within last 5 years.
19. Any other clinical condition that would jeopardize patients safety while participating in this clinical trial at the discretion of investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (56):
- China (38):
  - 1288.18.86001 Boehringer Ingelheim Investigational Site, Beijing
  - 1288.18.86002 Boehringer Ingelheim Investigational Site, Beijing
  - 1288.18.86003 Boehringer Ingelheim Investigational Site, Beijing
  - 1288.18.86004 Boehringer Ingelheim Investigational Site, Beijing
  - 1288.18.86046 Boehringer Ingelheim Investigational Site, Beijing
  - 1288.18.86019 Boehringer Ingelheim Investigational Site, Changchun
  - 1288.18.86020 Boehringer Ingelheim Investigational Site, Changchun
  - 1288.18.86028 Boehringer Ingelheim Investigational Site, Changsha
  - 1288.18.86029 Boehringer Ingelheim Investigational Site, Changsha
  - 1288.18.86050 Boehringer Ingelheim Investigational Site, Changsha
  - 1288.18.86045 Boehringer Ingelheim Investigational Site, Chengdu
  - 1288.18.86042 Boehringer Ingelheim Investigational Site, Chongqing
  - 1288.18.86023 Boehringer Ingelheim Investigational Site, Dalian
  - 1288.18.86009 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1288.18.86010 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1288.18.86012 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1288.18.86047 Boehringer Ingelheim Investigational Site, Haerbin
  - 1288.18.86032 Boehringer Ingelheim Investigational Site, Hefei
  - 1288.18.86016 Boehringer Ingelheim Investigational Site, Hengshui
  - 1288.18.86017 Boehringer Ingelheim Investigational Site, Jinan
  - 1288.18.86026 Boehringer Ingelheim Investigational Site, Lanzhou
  - 1288.18.86039 Boehringer Ingelheim Investigational Site, Nanchang
  - 1288.18.86035 Boehringer Ingelheim Investigational Site, Nanjing
  - 1288.18.86036 Boehringer Ingelheim Investigational Site, Nanjing
  - 1288.18.86034 Boehringer Ingelheim Investigational Site, Nanning
  - 1288.18.86006 Boehringer Ingelheim Investigational Site, Shanghai
  - 1288.18.86007 Boehringer Ingelheim Investigational Site, Shanghai
  - 1288.18.86008 Boehringer Ingelheim Investigational Site, Shanghai
  - 1288.18.86013 Boehringer Ingelheim Investigational Site, Shantou
  - 1288.18.86022 Boehringer Ingelheim Investigational Site, Shenyang
  - 1288.18.86014 Boehringer Ingelheim Investigational Site, Shijiazhuang
  - 1288.18.86015 Boehringer Ingelheim Investigational Site, Shijiazhuang
  - 1288.18.86038 Boehringer Ingelheim Investigational Site, Suzhou
  - 1288.18.86049 Boehringer Ingelheim Investigational Site, Wuhan
  - 1288.18.86033 Boehringer Ingelheim Investigational Site, Wuhu
  - 1288.18.86024 Boehringer Ingelheim Investigational Site, Xi'an
  - 1288.18.86025 Boehringer Ingelheim Investigational Site, Xi'an
  - 1288.18.86030 Boehringer Ingelheim Investigational Site, Yueyang
- Malaysia (8):
  - 1288.18.60004 Boehringer Ingelheim Investigational Site, Kelantan
  - 1288.18.60003 Boehringer Ingelheim Investigational Site, Kuala Selangor
  - 1288.18.60002 Boehringer Ingelheim Investigational Site, Malacca
  - 1288.18.60005 Boehringer Ingelheim Investigational Site, Negeri Sembilan
  - 1288.18.60007 Boehringer Ingelheim Investigational Site, Negeri Sembilan
  - 1288.18.60001 Boehringer Ingelheim Investigational Site, Perak
  - 1288.18.60006 Boehringer Ingelheim Investigational Site, Perak
  - 1288.18.60008 Boehringer Ingelheim Investigational Site, Putrajaya
- Philippines (7):
  - 1288.18.63007 Boehringer Ingelheim Investigational Site, Cebu
  - 1288.18.63003 Boehringer Ingelheim Investigational Site, Cebu City
  - 1288.18.63002 Boehringer Ingelheim Investigational Site, Makati City
  - 1288.18.63001 Boehringer Ingelheim Investigational Site, Manila
  - 1288.18.63008 Boehringer Ingelheim Investigational Site, Quezon City
  - 1288.18.63006 Boehringer Ingelheim Investigational Site, Surigao City
  - 1288.18.63005 Boehringer Ingelheim Investigational Site, Tagum
- Vietnam (3):
  - 1288.18.84003 Boehringer Ingelheim Investigational Site, Hanoi
  - 1288.18.84001 Boehringer Ingelheim Investigational Site, Ho Chi Minh City
  - 1288.18.84002 Boehringer Ingelheim Investigational Site, Ho Chi Minh City

REFERENCES:
- [Derived] Lv Q, Shen J, Miao L, Ye B, Schepers C, Plat A, Shi Y. Early Combination Therapy with Linagliptin and Metformin in People with Type 2 Diabetes Improves Glycemic Control to HbA1c </= 6.5% without Increasing Hypoglycemia: Pooled Analysis of Two Randomized Clinical Trials. Diabetes Ther. 2020 Jun;11(6):1317-1330. doi: 10.1007/s13300-020-00819-9. Epub 2020 Apr 23. PMID 32328953

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After 2-weeks placebo run-in in the main group, 730 of 733 randomised patients were treated in a double-blind fashion for 24 weeks. In the additional parallel group (APG), all of 143 randomised patients with HbA1c >=11% were treated for 24 weeks (the first 12 weeks were double-blind). There was a 1-week follow-up period after treatment.
Groups:
- Main: Linagliptin 5mg QD: Main Group: Patients received linagliptin 5mg once daily (QD), administered oral as tablet.
- Main: Metformin 500mg BID: Main Group: Patients received metformin 500mg twice daily (BID), administered oral as tablet.
- Main: Metformin 1000mg BID: Main Group: Patients received metformin 1000mg twice daily (BID), administered oral as tablet.
- Main: Linagliptin 2.5mg / Metformin 500mg BID: Main Group: Patients received linagliptin 2.5mg and metformin 500mg twice daily (BID), administered oral as fixed dose combination (FDC) tablet.
- Main: Linagliptin 2.5mg / Metformin 1000mg BID: Main Group: Patients received linagliptin 2.5mg and metformin 1000mg twice daily (BID), administered oral as fixed dose combination (FDC) tablet.
- APG: Linagliptin 5mg QD: Additional parallel group (APG): Patients received linagliptin 5mg once daily (QD), administered oral as tablet.
  (Data up to week 12)
- APG: Linagliptin 2.5mg / Metformin 1000mg BID: Additional parallel group (APG): Patients received linagliptin 2.5mg and metformin 1000mg twice daily (BID), administered oral as fixed dose combination (FDC) tablet.
  (Data up to week 12)
Period: Overall Study
Arm/Group | Main: Linagliptin 5mg QD | Main: Metformin 500mg BID | Main: Metformin 1000mg BID | Main: Linagliptin 2.5mg / Metformin 500mg BID | Main: Linagliptin 2.5mg / Metformin 1000mg BID | APG: Linagliptin 5mg QD | APG: Linagliptin 2.5mg / Metformin 1000mg BID
Started | 147 | 145 | 144 | 147 | 147 | 71 | 72
Completed | 130 | 137 | 127 | 137 | 131 | 64 | 65
Not Completed | 17 | 8 | 17 | 10 | 16 | 7 | 7
Not completed — Adverse Event | 3 | 4 | 9 | 2 | 7 | 3 | 5
Not completed — Lack of Efficacy | 3 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Non compliance with protocol | 0 | 2 | 1 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 2 | 2 | 0 | 0 | 1
Not completed — Refused to continue trial medication | 8 | 0 | 4 | 2 | 8 | 1 | 1
Not completed — Other Reason | 1 | 0 | 1 | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all patients treated with at least 1 dose of study medication
Groups:
- Main: Linagliptin 5mg QD: Main Group: Patients received linagliptin 5mg QD, administered oral as tablet.
- Main: Metformin 500mg BID: Main Group: Patients received metformin 500mg BID, administered oral as tablet.
- Main: Metformin 1000mg BID: Main Group: Patients received metformin 1000mg BID, administered oral as tablet.
- Main: Linagliptin 2.5mg / Metformin 500mg BID: Main Group: Patients received linagliptin 2.5mg and metformin 500mg BID, administered oral as fixed dose combination (FDC) tablet.
- Main: Linagliptin 2.5mg / Metformin 1000mg BID: Main Group: Patients received linagliptin 2.5mg and metformin 1000mg BID, administered oral as fixed dose combination (FDC) tablet.
- APG: Linagliptin 5mg QD: Additional parallel group (APG): Patients received linagliptin 5mg QD, administered oral as tablet.
  (Data up to week 12)
- APG: Linagliptin 2.5mg / Metformin 1000mg BID: Additional parallel group (APG): Patients received linagliptin 2.5mg and metformin 1000mg BID, administered oral as fixed dose combination (FDC) tablet.
  (Data up to week 12)
- Total: Total of all reporting groups
Arm/Group | Main: Linagliptin 5mg QD | Main: Metformin 500mg BID | Main: Metformin 1000mg BID | Main: Linagliptin 2.5mg / Metformin 500mg BID | Main: Linagliptin 2.5mg / Metformin 1000mg BID | APG: Linagliptin 5mg QD | APG: Linagliptin 2.5mg / Metformin 1000mg BID | Total
Number analyzed (Participants) | 147 | 145 | 144 | 147 | 147 | 71 | 72 | 873
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (10.5) | 52.1 (9.6) | 51.4 (10.4) | 51.4 (10.2) | 50.7 (9.4) | 49.5 (11.6) | 49.9 (11.7) | 51.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 54 | 53 | 55 | 60 | 23 | 32 | 348
  Male | 76 | 91 | 91 | 92 | 87 | 48 | 40 | 525

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in HbA1c After 24 Weeks of Treatment in Main Group
Description: The change from baseline in HbA1c after 24 weeks of treatment in main group.
  The mean was adjusted by baseline HbA1c and treatment group.
Time Frame: Baseline and week 24
Population: Full analysis set (FAS): all randomised and treated patients who had a baseline and at least 1 on-treatment HbA1c value As the imputation rule for missing data the last observation carried forward (LOCF) was used.
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Main: Linagliptin 5mg QD | Main: Metformin 500mg BID | Main: Metformin 1000mg BID | Main: Linagliptin 2.5mg / Metformin 500mg BID | Main: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 141 | 144 | 133 | 142 | 141
percentage | -1.29 (0.08) | -1.64 (0.08) | -2.07 (0.08) | -2.15 (0.08) | -2.29 (0.08)
Statistical Analysis 1: Comparison: Main: Metformin 1000mg BID vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; The model includes treatment as a fixed effect and baseline HbA1c as a linear covariate. The null and alternative hypotheses were tested in a hierarchical sequence. The next null hypothesis was tested in a confirmatory way only if all prior null-hypotheses were rejected. 'Greater effect' refers to a greater reduction in HbA1c; Test type: Superiority or Other; p = 0.0587, ANCOVA; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.45 to 0.01], Standard Error of Mean 0.12 — The adjusted mean difference was calculated as the adjusted mean of 'Main: Linagliptin 2.5mg / Metformin 1000mg BID' minus 'Main: Metformin 1000mg BID'
Statistical Analysis 2: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-1.23 to -0.78], Standard Error of Mean 0.11 — The adjusted mean difference was calculated as the adjusted mean of 'Main: Linagliptin 2.5mg / Metformin 1000mg BID' minus 'Main: Linagliptin 5mg QD'
Statistical Analysis 3: Comparison: Main: Metformin 500mg BID vs Main: Linagliptin 2.5mg / Metformin 500mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.73 to -0.29], Standard Error of Mean 0.11 — The adjusted mean difference was calculated as the adjusted mean of 'Main: Linagliptin 2.5mg / Metformin 500mg BID' minus 'Main: Metformin 500mg BID'
Statistical Analysis 4: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 500mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-1.09 to -0.64], Standard Error of Mean 0.11 — The adjusted mean difference was calculated as the adjusted mean of 'Main: Linagliptin 2.5mg / Metformin 500mg BID' minus 'Main: Linagliptin 5mg QD'

2. Secondary Outcome: The Occurrence of Treat to Target Efficacy Response in Terms of HbA1c < 7.0 % After 24 Weeks of Treatment in Main Group
Description: The occurrence of treat to target efficacy response in terms of HbA1c < 7.0 % after 24 weeks of treatment in main group.
Time Frame: Week 24 (after first drug administration)
Population: FAS - non-completers were considered as nonresponders (NCF)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main: Linagliptin 5mg QD | Main: Metformin 500mg BID | Main: Metformin 1000mg BID | Main: Linagliptin 2.5mg / Metformin 500mg BID | Main: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 140 | 144 | 129 | 140 | 140
percentage of participants | 43.6 [35.2 to 52.2] | 50.0 [41.6 to 58.4] | 69.0 [60.3 to 76.8] | 72.1 [63.9 to 79.4] | 77.1 [69.3 to 83.8]
Statistical Analysis 1: Comparison: Main: Metformin 1000mg BID vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; Comparison of 'Main: Linagliptin 2.5mg / Metformin 1000mg BID' / 'Main: Metformin 1000mg BID'. The logistic regression includes treatment and continuous baseline HbA1c; Test type: Superiority or Other; p = 0.0771, Regression, Logistic; Odds Ratio (OR) = 1.673, 95% CI 2-sided [0.946 to 2.961], Standard Error of Mean 0.487
Statistical Analysis 2: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; Comparison of 'Main: Linagliptin 2.5mg / Metformin 1000mg BID' / 'Main: Linagliptin 5mg QD'. The logistic regression includes treatment and continuous baseline HbA1c; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 5.489, 95% CI 2-sided [3.164 to 9.522], Standard Error of Mean 1.543
Statistical Analysis 3: Comparison: Main: Metformin 500mg BID vs Main: Linagliptin 2.5mg / Metformin 500mg BID; Comparison of 'Main: Linagliptin 2.5mg / Metformin 500mg BID' / 'Main: Metformin 500mg BID'. The logistic regression includes treatment and continuous baseline HbA1c; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.829, 95% CI 2-sided [1.678 to 4.767], Standard Error of Mean 0.753
Statistical Analysis 4: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 500mg BID; Comparison of 'Main: Linagliptin 2.5mg / Metformin 500mg BID' / 'Main: Linagliptin 5mg QD'. The logistic regression includes treatment and continuous baseline HbA1c; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.818, 95% CI 2-sided [2.259 to 6.454], Standard Error of Mean 1.023

3. Secondary Outcome: The Occurrence of Treat to Target Efficacy Response in Terms of HbA1c < 7.0 % After 12 Weeks of Treatment in APG
Description: The occurrence of treat to target efficacy response in terms of HbA1c < 7.0 % after 12 weeks of treatment in APG.
Time Frame: Week 12 (after first drug administration)
Population: FAS (NCF)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | APG: Linagliptin 5mg QD | APG: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 70 | 68
percentage of participants | 27.1 [17.2 to 39.1] | 58.8 [46.2 to 70.6]
Statistical Analysis 1: Comparison: APG: Linagliptin 5mg QD vs APG: Linagliptin 2.5mg / Metformin 1000mg BID; Comparison of 'APG: Linagliptin 2.5mg / Metformin 1000mg BID' / 'APG: Linagliptin 5mg QD'. The logistic regression includes treatment and continuous baseline HbA1c; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.169, 95% CI 2-sided [1.997 to 8.701], Standard Error of Mean 1.565

4. Secondary Outcome: The Occurrence of Treat to Target Efficacy Response in Terms of HbA1c < 6.5% After 24 Weeks of Treatment in Main Group
Description: The occurrence of treat to target efficacy response in terms of HbA1c < 6.5% after 24 weeks of treatment in main group.
Time Frame: Week 24 (after first drug administration)
Population: FAS (NCF)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main: Linagliptin 5mg QD | Main: Metformin 500mg BID | Main: Metformin 1000mg BID | Main: Linagliptin 2.5mg / Metformin 500mg BID | Main: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 141 | 144 | 133 | 142 | 141
percentage of participants | 23.4 [16.7 to 31.3] | 34.7 [27.0 to 43.1] | 50.4 [41.6 to 59.2] | 56.3 [47.8 to 64.6] | 60.3 [51.7 to 68.4]
Statistical Analysis 1: Comparison: Main: Metformin 1000mg BID vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0480, Regression, Logistic; Odds Ratio (OR) = 1.661, 95% CI 2-sided [1.004 to 2.746], Standard Error of Mean 0.426
Statistical Analysis 2: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 5.923, 95% CI 2-sided [3.452 to 10.164], Standard Error of Mean 1.632
Statistical Analysis 3: Comparison: Main: Metformin 500mg BID vs Main: Linagliptin 2.5mg / Metformin 500mg BID; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 2.574, 95% CI 2-sided [1.563 to 4.239], Standard Error of Mean 0.655
Statistical Analysis 4: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 500mg BID; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.682, 95% CI 2-sided [2.751 to 7.968], Standard Error of Mean 1.270

5. Secondary Outcome: The Occurrence of Treat to Target Efficacy Response in Terms of HbA1c < 6.5% After 12 Weeks of Treatment in APG
Description: The occurrence of treat to target efficacy response in terms of HbA1c < 6.5% after 12 weeks of treatment in APG.
Time Frame: Week 12 (after first drug administration)
Population: FAS (NCF)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | APG: Linagliptin 5mg QD | APG: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 70 | 68
percentage of participants | 15.7 [8.1 to 26.4] | 36.8 [25.4 to 49.3]
Statistical Analysis 1: Comparison: APG: Linagliptin 5mg QD vs APG: Linagliptin 2.5mg / Metformin 1000mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0062, Regression, Logistic; Odds Ratio (OR) = 3.135, 95% CI 2-sided [1.383 to 7.110], Standard Error of Mean 1.310

6. Primary Outcome: The Change From Baseline in HbA1c After 24 Weeks of Treatment in Main Group - FAS (OC)
Description: The change from baseline in HbA1c after 24 weeks of treatment in main group. Only subjects from the FAS with measured HbA1c values (observed cases [OC]) were considered.
  The mean was adjusted by treatment, baseline HbA1c, week and treatment*week.
  The sensitivity analysis was added as the primary analysis failed with borderline results.
Time Frame: Baseline and week 24
Population: FAS (OC): subjects from the FAS with measured HbA1c values (observed cases [OC]) were considered
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Main: Linagliptin 5mg QD | Main: Metformin 500mg BID | Main: Metformin 1000mg BID | Main: Linagliptin 2.5mg / Metformin 500mg BID | Main: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 125 | 133 | 127 | 135 | 128
percentage | -1.34 (0.08) | -1.68 (0.08) | -2.08 (0.08) | -2.16 (0.08) | -2.38 (0.08)
Statistical Analysis 1: Comparison: Main: Metformin 1000mg BID vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; Sensitivity analysis: Mixed Model for repeated measurements The model includes baseline HbA1c as a linear covariate; visit, treatment and visit by treatment interaction as fixed classification effects and patient as a random effect with unstructured covariance structure to model within-patients errors; Test type: Superiority or Other; p = 0.0109, ANCOVA; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.53 to -0.07], Standard Error of Mean 0.12 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-1.27 to -0.81], Standard Error of Mean 0.12 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Main: Metformin 500mg BID vs Main: Linagliptin 2.5mg / Metformin 500mg BID; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.70 to -0.24], Standard Error of Mean 0.12 — The adjusted mean difference was calculated as the adjusted mean of 'Main: Linagliptin 2.5mg / Metformin 500mg BID ' minus 'Main: Metformin 500mg BID'
Statistical Analysis 4: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 500mg BID; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.04 to -0.58], Standard Error of Mean 0.12 — [estimate comment as in outcome 1, analysis 4]

7. Primary Outcome: The Change From Baseline in HbA1c After 12 Weeks of Treatment in APG
Description: The change from baseline in HbA1c after 12 weeks of treatment in additional parallel group (APG)
  The mean was adjusted by baseline HbA1c and treatment group.
Time Frame: Baseline and week 12
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: percentage
Arm/Group | APG: Linagliptin 5mg QD | APG: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 70 | 68
percentage | -3.46 (0.22) | -4.71 (0.22)
Statistical Analysis 1: Comparison: APG: Linagliptin 5mg QD vs APG: Linagliptin 2.5mg / Metformin 1000mg BID; The treatment effect of the 'APG: Linagliptin 2.5mg / Metformin 1000mg BID' was compared with 'APG: Linagliptin 5mg QD'. The model includes treatment as a fixed effect and baseline HbA1c as a linear covariate; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-1.87 to -0.63], Standard Error of Mean 0.32 — The adjusted mean difference was calculated as the adjusted mean of 'APG: Linagliptin 2.5mg / Metformin 1000mg BID' minus 'APG: Linagliptin 5mg QD'

8. Secondary Outcome: The Occurrence of Relative Efficacy Response in Main Group
Description: The occurrence of relative efficacy response (HbA1c lowering by at least 0.5% after 24 weeks of treatment) in main group
Time Frame: From baseline until week 24
Population: FAS (NCF)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main: Linagliptin 5mg QD | Main: Metformin 500mg BID | Main: Metformin 1000mg BID | Main: Linagliptin 2.5mg / Metformin 500mg BID | Main: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 141 | 144 | 133 | 142 | 141
percentage of participants | 73.0 [64.9 to 80.2] | 80.6 [73.1 to 86.7] | 89.5 [83.0 to 94.1] | 93.0 [87.4 to 96.6] | 89.4 [83.1 to 93.9]
Statistical Analysis 1: Comparison: Main: Metformin 1000mg BID vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9705, Regression, Logistic; Odds Ratio (OR) = 0.986, 95% CI 2-sided [0.456 to 2.130], Standard Error of Mean 0.387
Statistical Analysis 2: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 3.093, 95% CI 2-sided [1.612 to 5.938], Standard Error of Mean 1.029
Statistical Analysis 3: Comparison: Main: Metformin 500mg BID vs Main: Linagliptin 2.5mg / Metformin 500mg BID; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0029, Regression, Logistic; Odds Ratio (OR) = 3.190, 95% CI 2-sided [1.486 to 6.849], Standard Error of Mean 1.243
Statistical Analysis 4: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 500mg BID; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.871, 95% CI 2-sided [2.318 to 10.238], Standard Error of Mean 1.846

9. Secondary Outcome: The Occurrence of Relative Efficacy Response in APG
Description: The Occurrence of Relative Efficacy Response (HbA1c Lowering by at Least 0.5% After 12 Weeks of Treatment) in APG
Time Frame: From baseline until week 12
Population: FAS (NCF)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | APG: Linagliptin 5mg QD | APG: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 70 | 68
percentage of participants | 84.3 [73.6 to 91.9] | 91.2 [81.8 to 96.7]
Statistical Analysis 1: Comparison: APG: Linagliptin 5mg QD vs APG: Linagliptin 2.5mg / Metformin 1000mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2523, Regression, Logistic; Odds Ratio (OR) = 1.865, 95% CI 2-sided [0.642 to 5.420], Standard Error of Mean 1.015

10. Secondary Outcome: The Change in Fasting Plasma Glucose (FPG) From Baseline After 24 Weeks of Treatment in Main Group
Description: The change in fasting plasma glucose (FPG) from baseline after 24 weeks of treatment in main group.
  Adjusted mean: The model includes continuous baseline HbA1c, continuous baseline FPG and treatment group.
Time Frame: Baseline and week 24
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Main: Linagliptin 5mg QD | Main: Metformin 500mg BID | Main: Metformin 1000mg BID | Main: Linagliptin 2.5mg / Metformin 500mg BID | Main: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 140 | 144 | 133 | 142 | 140
mg/dL | -15.03 (2.25) | -29.87 (2.23) | -42.07 (2.31) | -39.33 (2.24) | -47.44 (2.26)
Statistical Analysis 1: Comparison: Main: Metformin 1000mg BID vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; The model includes continuous baseline HbA1c, continuous baseline FPG and treatment group; Test type: Superiority or Other; p = 0.0971, ANCOVA; Mean Difference (Final Values) = -5.37, 95% CI 2-sided [-11.72 to 0.98], Standard Error of Mean 3.23 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; The model includes continuous baseline HbA1c, continuous baseline FPG and treatment group; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -32.42, 95% CI 2-sided [-38.67 to -26.16], Standard Error of Mean 3.19 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Main: Metformin 500mg BID vs Main: Linagliptin 2.5mg / Metformin 500mg BID; The model includes continuous baseline HbA1c, continuous baseline FPG and treatment group; Test type: Superiority or Other; p = 0.0028, ANCOVA; Median Difference (Net) = -9.47, 95% CI 2-sided [-15.66 to -3.27], Standard Error of Mean 3.16 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 500mg BID; The model includes continuous baseline HbA1c, continuous baseline FPG and treatment group; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -24.31, 95% CI 2-sided [-30.54 to -18.08], Standard Error of Mean 3.17 — [estimate comment as in outcome 1, analysis 4]

11. Secondary Outcome: The Change in Fasting Plasma Glucose (FPG) From Baseline After 12 Weeks of Treatment in APG
Description: The Change in Fasting Plasma Glucose (FPG) From Baseline After 12 Weeks of Treatment in APG.
  Adjusted mean: The model includes continuous baseline HbA1c, continuous baseline FPG and treatment group.
Time Frame: Baseline and week 12
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | APG: Linagliptin 5mg QD | APG: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 66 | 67
mg/dL | -56.70 (6.53) | -91.92 (6.48)
Statistical Analysis 1: Comparison: APG: Linagliptin 5mg QD vs APG: Linagliptin 2.5mg / Metformin 1000mg BID; The model includes continuous baseline HbA1c, continuous baseline FPG and treatment group; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -35.21, 95% CI 2-sided [-53.48 to -16.95], Standard Error of Mean 9.23 — [estimate comment as in outcome 7, analysis 1]

12. Secondary Outcome: The Frequency of Patients With Use of Rescue Therapy During 24 Week Treatment Period in Main Group
Description: The frequency of patients with use of rescue therapy during 24 week treatment period in main group.
  For this analysis the main group contrast 'Metformin 1000mg BID, Linagliptin 2.5mg / Metformin 1000mg BID' could not be analysed due to lack of events in the Metformin 1000mg BID group.
Time Frame: From baseline until week 24
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main: Linagliptin 5mg QD | Main: Metformin 500mg BID | Main: Metformin 1000mg BID | Main: Linagliptin 2.5mg / Metformin 500mg BID | Main: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 141 | 144 | 133 | 142 | 141
percentage of participants | 7.1 [3.5 to 12.7] | 2.1 [0.4 to 6.0] | 0.0 [0.0 to 2.7] | 1.4 [0.2 to 5.0] | 2.1 [0.4 to 6.1]
Statistical Analysis 1: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 1000mg BID; Comparison of 'Main: Linagliptin 2.5mg / Metformin 1000mg BID' / 'Main: Linagliptin 5mg QD'. The logistic regression includes treatment and continuous baseline HbA1c. The validity of the model is questionable as there is possibly a quasi-complete separation of data points, the results shown are based on the last maximum likelihood iteration; Test type: Superiority or Other; p = 0.0271, Regression, Logistic; Odds Ratio (OR) = 0.209, 95% CI 2-sided [0.052 to 0.838], Standard Error of Mean 0.148
Statistical Analysis 2: Comparison: Main: Metformin 500mg BID vs Main: Linagliptin 2.5mg / Metformin 500mg BID; Comparison of 'Main: Linagliptin 2.5mg / Metformin 500mg BID' / 'Main: Metformin 500mg BID'. The logistic regression includes treatment and continuous baseline HbA1c. The validity of the model is questionable as there is possibly a quasi-complete separation of data points, the results shown are based on the last maximum likelihood iteration; Test type: Superiority or Other; p = 0.9699, Regression, Logistic; Odds Ratio (OR) = 0.965, 95% CI 2-sided [0.150 to 6.202], Standard Error of Mean 0.916
Statistical Analysis 3: Comparison: Main: Linagliptin 5mg QD vs Main: Linagliptin 2.5mg / Metformin 500mg BID; Comparison of 'Main: Linagliptin 2.5mg / Metformin 500mg BID' / 'Main: Linagliptin 5mg QD'. The logistic regression includes treatment and continuous baseline HbA1c. The validity of the model is questionable as there is possibly a quasi-complete separation of data points, the results shown are based on the last maximum likelihood iteration; Test type: Superiority or Other; p = 0.0343, Regression, Logistic; Odds Ratio (OR) = 0.183, 95% CI 2-sided [0.038 to 0.882], Standard Error of Mean 0.147

13. Secondary Outcome: The Frequency of Patients With Use of Rescue Therapy During 12 Week Treatment Period in APG
Description: The Frequency of Patients With Use of Rescue Therapy During 12 Week Treatment Period in APG.
Time Frame: From baseline until week 12
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | APG: Linagliptin 5mg QD | APG: Linagliptin 2.5mg / Metformin 1000mg BID
Number analyzed (Participants) | 70 | 68
percentage of participants | 10.0 [4.1 to 19.5] | 1.5 [0.0 to 7.9]
Statistical Analysis 1: Comparison: APG: Linagliptin 5mg QD vs APG: Linagliptin 2.5mg / Metformin 1000mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0474, Regression, Logistic; Odds Ratio (OR) = 0.114, 95% CI 2-sided [0.013 to 0.976], Standard Error of Mean 0.125

ADVERSE EVENTS:
Time Frame: From first drug administration (week 1) until end of treatment, up to 24 weeks
Groups:
- Main: Linagliptin 5mg QD: Main Group: Patients once daily received linagliptin 5mg QD, administered oral as tablet.
- Main: Metformin 500mg BID: Main Group: Patients twice daily received metformin 500mg BID, administered oral as tablet.
- Main: Metformin 1000mg BID: Main Group: Patients twice daily received metformin 1000mg BID, administered oral as tablet.
- Main: Linagliptin 2.5mg / Metformin 500mg BID: Main Group: Patients twice daily received linagliptin 2.5mg and metformin 500mg BID, administered oral as fixed dose combination (FDC) tablet.
- Main: Linagliptin 2.5mg / Metformin 1000mg BID: Main Group: Patients twice daily received linagliptin 2.5mg and metformin 1000mg BID, administered oral as fixed dose combination (FDC) tablet.
- APG: Linagliptin 5mg QD up to Week 12: Additional parallel group (APG): Patients once daily received linagliptin 5mg QD, administered oral as tablet.
  (Data up to week 12)
- APG: Linagliptin 2.5mg / Metformin 1000mg BID up to Week 12: Additional parallel group (APG): Patients twice daily received linagliptin 2.5mg and metformin 1000mg BID, administered oral as fixed dose combination (FDC) tablet.
  (Data up to week 12)
- APG: Linagliptin 5mg After Week 12: Additional parallel group (APG): Patients once daily received linagliptin 5mg QD, administered oral as tablet. Data from week 12 to week 24
- APG: Linagliptin 5mg - Linagliptin 2.5mg / Met After Week 12: Additional parallel group (APG): Patients who received linagliptin 5mg QD, administered oral as tablet during the first 12 weeks and switched to linagliptin 2.5mg and metformin 1000mg (met) BID, administered oral as fixed dose combination (FDC) tablet from week 12 to week 24. Data from week 12 to week 24.
- APG: Linagliptin 2.5mg / Metformin 1000mg After Week 12: Additional parallel group (APG): Patients twice daily received linagliptin 2.5mg and metformin 1000mg BID, administered oral as fixed dose combination (FDC) tablet.
  Data from week 12 to week 24.
Arm/Group | Main: Linagliptin 5mg QD | Main: Metformin 500mg BID | Main: Metformin 1000mg BID | Main: Linagliptin 2.5mg / Metformin 500mg BID | Main: Linagliptin 2.5mg / Metformin 1000mg BID | APG: Linagliptin 5mg QD up to Week 12 | APG: Linagliptin 2.5mg / Metformin 1000mg BID up to Week 12 | APG: Linagliptin 5mg After Week 12 | APG: Linagliptin 5mg - Linagliptin 2.5mg / Met After Week 12 | APG: Linagliptin 2.5mg / Metformin 1000mg After Week 12
Serious Adverse Events (participants affected / at risk) | 2/147 | 1/145 | 2/144 | 1/147 | 4/147 | 1/71 | 1/72 | 0/33 | 1/31 | 1/65
Other Adverse Events (participants affected / at risk) | 30/147 | 31/145 | 42/144 | 32/147 | 41/147 | 20/71 | 15/72 | 2/33 | 9/31 | 9/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main: Linagliptin 5mg QD (N=147) | Main: Metformin 500mg BID (N=145) | Main: Metformin 1000mg BID (N=144) | Main: Linagliptin 2.5mg / Metformin 500mg BID (N=147) | Main: Linagliptin 2.5mg / Metformin 1000mg BID (N=147) | APG: Linagliptin 5mg QD up to Week 12 (N=71) | APG: Linagliptin 2.5mg / Metformin 1000mg BID up to Week 12 (N=72) | APG: Linagliptin 5mg After Week 12 (N=33) | APG: Linagliptin 5mg - Linagliptin 2.5mg / Met After Week 12 (N=31) | APG: Linagliptin 2.5mg / Metformin 1000mg After Week 12 (N=65)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otosclerosis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main: Linagliptin 5mg QD (N=147) | Main: Metformin 500mg BID (N=145) | Main: Metformin 1000mg BID (N=144) | Main: Linagliptin 2.5mg / Metformin 500mg BID (N=147) | Main: Linagliptin 2.5mg / Metformin 1000mg BID (N=147) | APG: Linagliptin 5mg QD up to Week 12 (N=71) | APG: Linagliptin 2.5mg / Metformin 1000mg BID up to Week 12 (N=72) | APG: Linagliptin 5mg After Week 12 (N=33) | APG: Linagliptin 5mg - Linagliptin 2.5mg / Met After Week 12 (N=31) | APG: Linagliptin 2.5mg / Metformin 1000mg After Week 12 (N=65)
Upper respiratory tract infection (Infections and infestations) | 6 | 6 | 14 | 12 | 11 | 2 | 4 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 3 | 2 | 4 | 4 | 2 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 4 | 0 | 4 | 2 | 12 | 2 | 0 | 2 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 13 | 13 | 8 | 11 | 4 | 4 | 1 | 6 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 3 | 4 | 5 | 10 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 8 | 16 | 7 | 14 | 2 | 4 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 2 | 7 | 3 | 6 | 1 | 2 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.